CLINICAL TRIAL: NCT05634213
Title: Feasibility of Transepicardial Atrial Injection of Saline at the Time Open Chest Cardiac Surgery
Brief Title: Feasibility of Transepicardial Atrial Injection
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Logistical issues
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pending
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- saline injection (Experimental): After the patient is placed on cardiopulmonary bypass, the surgeon will inject a saline into the atria.
  Interventions: Drug: normal saline
- standard of care (No Intervention): The patient will be placed on cardiopulmonary bypass as usual and the surgery will proceed without an attempt to inject saline into the atrial tissue.

INTERVENTIONS:
Drug: normal saline — Once the patient is placed on cardiopulmonary bypass, the product will be injected into the left atrial wall using a 27 gauge needle as 4 injections of 200 μL each. Two will be placed in the atrial appendage. The remaining 2 injections will be placed equidistant on the anterior atrial free wall. Each injection will be performed just under the surface of the atrial epicardium over 30 seconds. The needle will stay in place for 10 seconds after the injection to limit back flow from the site of injection.
  Other Names: 0.9% sodium chloride
  Arms: saline injection

SUMMARY:
Single blind feasibility trial using a binary 'traffic light' design to evaluate the feasibility of injecting normal physiological saline into the atria of patients at the time of clinically indicated open chest cardiac surgery.

DETAILED DESCRIPTION:
In this project, The investigators will see if patients can undergo successful transepicardial injection of saline at the time of cardiac surgery as compared to no injection. Patients will be randomised in a 1:1 allocation ratio using a parallel two-arm design. The study is designed to meet the following 3 feasibility objectives before proceeding: reasonable recruitment uptake, successful transepicardial injection of saline into the atria, and adequate retention of patients at follow-up.

ELIGIBILITY:
Inclusion Criteria:

Undergoing non-emergent open chest cardiac surgery for coronary artery bypass graft (CABG) and/or valve disease.

Exclusion Criteria:

1. Age less than or equal to 18 years of age.
2. Pregnant or breast feeding.
3. Patient is unable or unwilling to provide informed consent.
4. Patient is included in another randomized clinical trial.
5. A history of complex congenital heart disease.
6. Presence of any active malignancy (other than non-melanoma skin cancer) that required treatment within the last 2 years.
7. Underwent ineligible procedures during or prior to operation (including atrial ﬁbrillation ablation, heart transplantation, pulmonary thromboendarterectomy, isolated thoracic aorta procedures, ventricular assist device insertion, extracorporeal membrane oxygenator insertion, and percutaneous valve replacement).
8. Patients for whom the investigator believes that the trial is not in the interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment uptake | 1 year
  Recruitment uptake <20% (project not feasible), 20-35% (protocol needs to be revised), and > 35% (project feasible).
Treatment fidelity | 1 year
  Treatment successfully applied < 50% (approach not feasible), 50-75% (approach needs to be revised) and > 75% (approach is feasible).
Participant retention (follow up) | 30 days post surgery
  Follow up: < 65% (project not feasible), 65-85% (follow-up needs to be revised), > 85% (project is feasible).

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Davis, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Insitute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No